CLINICAL TRIAL: NCT06362252
Title: A Phase 1b/2, Multicenter, Open-label Study of Ifinatamab Deruxtecan (I-DXd), a B7-H3 Antibody-Drug Conjugate (ADC), in Combination With Atezolizumab With or Without Carboplatin as First-line Induction or Maintenance, in Subjects With Extensive-stage Small Cell Lung Cancer (ES-SCLC) (IDeate-Lung03)
Brief Title: A Study of I-DXd in Combination With Atezolizumab With or Without Carboplatin as First-Line Induction or Maintenance in Subjects With Extensive Stage-Small Cell Lung Cancer (IDeate-Lung03)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS7300-189; 2023-509629-36 (Other: EU CT); 2031240089 (Other: JRCT)
Record Dates: First submitted 2024-01-02; First posted 2024-04-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Extensive Stage-small Cell Lung Cancer
Keywords: Extensive stage-small cell lung cancer (ES-SCLC); Ifinatamab deruxtecan; I-DXd
MeSH Terms: interventions — atezolizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1, Part A: Maintenance Only (I-DXd 12 mg/kg) (Experimental): Part A (Safety Run-in): Participants who must have received 4 cycles of 1L induction standard of care (SoC) therapy with best overall response of CR, PR, or SD will receive maintenance therapy only. Maintenance therapy consisting of I-DXd 12 mg/kg (or a lower dose based on data for I-DXd collected during the study) + atezolizumab 1200 mg IV Q3W.
  A 5-day surveillance period between each of the first 3 participants (up to a maximum of 9 participants) dosed is included as a safety measure.
  Interventions: Drug: Ifinatamab deruxtecan; Drug: Atezolizumab
- Cohort 2, Part A: Induction + Maintenance (I-DXd 8 mg/kg) (Experimental): Part A (Safety Run-in): Participants who are treatment-naive, newly diagnosed with ES-SCLC will receive 4 cycles of 1L I-DXd induction therapy (8 mg/kg IV Q3W) + atezolizumab (1200 mg IV Q3W) + carboplatin (AUC 5 mg/ml×min IV Q3W) followed by maintenance therapy. Maintenance therapy consisting of I-DXd 8 mg/kg (or a lower dose based on data for I-DXd collected during the study) + atezolizumab 1200 mg IV Q3W.
  Interventions: Drug: Ifinatamab deruxtecan; Drug: Atezolizumab; Drug: Carboplatin
- Cohort 2, Part A: Induction + Maintenance (I-DXd 12 mg/kg) (Experimental): Part A (Safety Run-in): Participants who are treatment-naive, newly diagnosed with ES-SCLC will receive 4 cycles of 1L I-DXd induction therapy (12 mg/kg IV Q3W) + atezolizumab (1200 mg IV Q3W) + carboplatin (AUC 5 mg/ml×min IV Q3W) followed by maintenance therapy. Maintenance therapy consisting of I-DXd 12 mg/kg (or a lower dose based on data for I-DXd collected during the study) + atezolizumab 1200 mg IV Q3W.
  Interventions: Drug: Ifinatamab deruxtecan; Drug: Atezolizumab; Drug: Carboplatin
- Cohort 1, Part B: Maintenance (I-DXd 8 mg/kg) (Experimental): Part B: Participants who must have received 4 cycles of 1L induction standard of care (SoC) therapy with best overall response of CR, PR, or SD will receive maintenance therapy only starting at Cycle 1 Day 1. Maintenance therapy consisting of I-DXd 8 mg/kg (or a lower dose based on data for I-DXd collected during the study) + atezolizumab 1200 mg IV Q3W
  Interventions: Drug: Ifinatamab deruxtecan; Drug: Atezolizumab
- Cohort 1, Part B: Maintenance (I-DXd 12 mg/kg) (Experimental): Part B: Participants who must have received 4 cycles of 1L induction standard of care (SoC) therapy with best overall response of CR, PR, or SD will receive maintenance therapy only starting at Cycle 1 Day 1. Maintenance therapy consisting of I-DXd 12 mg/kg (or a lower dose based on data for I-DXd collected during the study) + atezolizumab 1200 mg IV Q3W.
  Interventions: Drug: Ifinatamab deruxtecan; Drug: Atezolizumab
- Cohort 2, Part B: Induction + Maintenance (I-DXd 8 mg/kg) (Experimental): Participants who are treatment-naive, newly diagnosed with ES-SCLC will receive 4 cycles of 1L I-DXd induction therapy (8 mg/kg IV Q3W) + atezolizumab (1200 mg IV Q3W) + carboplatin (AUC 5 mg/ml×min IV Q3W) followed by maintenance therapy. Maintenance therapy consisting of I-DXd 8 mg/kg (or a lower dose based on data for I-DXd collected during the study) + atezolizumab 1200 mg IV Q3W.
  Interventions: Drug: Ifinatamab deruxtecan; Drug: Atezolizumab; Drug: Carboplatin
- Cohort 2, Part B: Induction + Maintenance (I-DXd 12 mg/kg) (Experimental): Participants who are treatment-naive, newly diagnosed with ES-SCLC will receive 4 cycles of IL I-DXd induction therapy (12 mg/kg IV Q3W) + atezolizumab (1200 mg IV Q3W) + carboplatin (AUC 5 mg/ml×minIV Q3W) followed by maintenance therapy. Maintenance therapy consisting of I-DXd 12 mg/kg (or a lower dose based on data for I-DXd collected during the study) + atezolizumab 1200 mg IV Q3W.
  Interventions: Drug: Ifinatamab deruxtecan; Drug: Atezolizumab; Drug: Carboplatin

INTERVENTIONS:
Drug: Ifinatamab deruxtecan — Intravenous administration
  Other Names: I-DXd
Drug: Atezolizumab — Intravenous administration
Drug: Carboplatin — Intravenous administration
  Arms: Cohort 2, Part A: Induction + Maintenance (I-DXd 12 mg/kg); Cohort 2, Part A: Induction + Maintenance (I-DXd 8 mg/kg); Cohort 2, Part B: Induction + Maintenance (I-DXd 12 mg/kg); Cohort 2, Part B: Induction + Maintenance (I-DXd 8 mg/kg)

SUMMARY:
This study is designed to evaluate the safety and efficacy of ifinatamab deruxtecan (I-DXd) in combination with immune checkpoint inhibitor (ICI) atezolizumab with or without carboplatin in participants with extensive stage-small cell lung cancer (ES-SCLC) in the first-line (1L) setting.

DETAILED DESCRIPTION:
This study consists of two parts and two cohorts: Part A (Phase 1b; Safety Run-in) and Part B (Phase 2; Dose Optimization), Cohort 1 (I-DXd in maintenance) and Cohort 2 (I-DXd in induction + maintenance).

The primary objective of this study is to evaluate the safety and tolerability of I-DXd in combination with atezolizumab with or without carboplatin by assessing treatment-emergent adverse events (TEAEs) and other safety parameters which will inform optimal dose selection of I-DXd in the combination regimens (Dose Optimization Part B) of this study.

ELIGIBILITY:
A full list of inclusion/exclusion criteria are available in the protocol.

Inclusion Criteria

Participants must meet all of the following criteria to be eligible for enrollment into the study:

1. Sign and date the informed consent form (ICF), prior to the start of any study-specific qualification procedures.
2. Adults ≥18 years or the minimum legal adult age (whichever is greater) at the time the ICF is signed.
3. Has histologically or cytologically confirmed diagnosis of ES-SCLC who will require first-line (IL) therapy.
4. For Cohort 1, participant has received 4 cycles of 1L induction therapy with carboplatin, etoposide, and atezolizumab for ES-SCLC with ongoing CR PR, CR, or SD per RECIST v1.1 assessed by the investigator.

   For Cohort 2, participant has received no prior treatment for ES-SCLC.
5. For Cohort 2, participant has at least one measurable lesion according to RECIST v1.1 on computed tomography (CT) or magnetic resonance imaging (MRI) as assessed by the investigator.
6. For Cohort 2, participant must have at least one lesion, amenable to core biopsy, and must consent to provide a pretreatment biopsy tissue sample and on-treatment biopsy.
7. Has ECOG PS of ≤1 (assessed within 7 days before enrollment/randomization).
8. Has adequate organ and bone marrow function within 7 days before the start of study treatment as specified in the study protocol.
9. A female subject of childbearing potential (POCBP) is eligible to participate if the following conditions are met:

   1. Subject is not pregnant as confirmed by highly sensitive pregnancy test during Screening (within 3 days prior to enrollment/randomization)
   2. Subject does not breastfeed during the treatment period and for at least 8/5/6 months after last dose of I-DXd/atezolizumab/carboplatin, respectively.
   3. Subject agrees to adhere to a contraceptive method that is highly effective and agrees not to donate eggs (ova, oocytes) to others or freeze/store eggs during the treatment period and for at least the time needed to eliminate each study drug after the last dose. The length of time required to continue contraception and avoid donating/freezing eggs after last dose for I-DXd/atezolizumab/carboplatin is 8/5/6 months, respectively. Preservation of eggs may be considered prior to first dose of study drug.
10. A male subject capable of producing sperm is eligible to participate if he agrees to the following during the intervention period and for at least the time needed to eliminate each study drug. The length of time required to continue contraception and avoid donating sperm after last dose for I-DXd/atezolizumab/carboplatin is 6/5/6 months, respectively.

    1. Avoid donating sperm.
    2. Adhere to either of the contraception methods: true abstinence from penile-vaginal intercourse or uses a penile/external condom when having penile-vaginal intercourse with a non-subject of childbearing potential plus partner use of an additional contraceptive method.
11. Is willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures, and study restrictions.

Exclusion Criteria

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Has received prior treatment with orlotamab, enoblituzumab, or other B7-H3 targeted agents, including I-DXd.
2. Prior discontinuation of an ADC that consists of an exatecan derivative (eg, trastuzumab deruxtecan) due to treatment-related toxicities.
3. Has received prior treatment with CD137 agonists or ICIs, including anti-cytotoxic T-cell lymphocyte-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, except for atezolizumab for Cohort 1.
4. Has inadequate washout period before enrollment/randomization as specified in the study protocol.
5. Has any of the following within the past 6 months: cerebrovascular accident, transient ischemic attack, or another arterial thromboembolic event.
6. Has clinically active brain metastases, spinal cord compression, or leptomeningeal carcinomatosis, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms.
7. Has clinically significant corneal disease.
8. Has uncontrolled or significant cardiovascular disease,.
9. Has history of (non-infectious) ILD/pneumonitis that required corticosteroids, current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at Screening.
10. Has clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
11. Is on chronic steroid treatment (dose of 10 mg daily or more prednisone equivalent), except for low-dose inhaled steroids (for asthma/chronic obstructive pulmonary disease, topical steroids (for mild skin conditions), or intra-articular steroid injections.
12. Has history of malignancy other than SCLC within the 5 years prior to randomization/enrollment, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, superficial gastrointestinal tract tumors, and non-muscle invasive bladder cancer curatively resected by endoscopic surgery.
13. Has history of allogeneic bone marrow, stem cell, or solid organ transplant.
14. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI-CTCAE V5.0, Grade ≤1 or baseline.
15. Has history of hypersensitivity to the drug substances, inactive ingredients in the drug product or severe hypersensitivity reactions to other monoclonal antibodies.
16. Has evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection.
17. Has active or uncontrolled human immunodeficiency virus (HIV) infection.
18. Has active or uncontrolled hepatitis B or C virus (HBV or HCV) infection.
19. Has history of autoimmune disease.
20. Has any evidence of severe or uncontrolled systemic diseases.
21. Has received a live vaccine within 30 days prior to the first dose of study drug.
22. Is a female who is pregnant or breastfeeding or planning to become pregnant.
23. Has prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the participant; alter the absorption, distribution, metabolism, or excretion of the study drug; or confound the assessment of study results.
24. Has psychological, social, familial, or logistical factors that would prevent regular follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Reporting Dose-limiting Toxicities Following I-DXd in Combination With Atezolizumab With or Without Carboplatin (Part A) | Cycle 1 Day 1 up to Cycle 1 Day 21 (each cycle is 21 days)
Overall Number of Participants With Treatment-emergent Adverse Events Following I-DXd in Combination With Atezolizumab With or Without Carboplatin (Part A and B) | Baseline up to 37 months

SECONDARY OUTCOMES:
Progression-free Survival As Assessed by Blinded Independent Central Review and Investigator Following I-DXd in Combination With Atezolizumab With or Without Carboplatin (Part A and B) | From start date of study drug to the earlier date of the first objective documentation of radiographic disease progression assessed by BICR and investigator per RECIST v1.1 or death due to any cause, whichever occurs first, up to approximately 37 months
  Progression-free survival is defined as the time from the enrollment/randomization date to the earlier of the dates of the first documentation of disease progression assessed by BICR and investigator per RECIST v1.1 or death due to any cause.
Objective Response Rate Assessed by Blinded Independent Central Review and Investigator Following I-DXd in Combination With Atezolizumab With Carboplatin (Part A and B of Cohort 2 Only) | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 37 months
  Objective response rate (ORR) is defined as proportion of subjects who achieved a best overall response of confirmed complete response (CR) or confirmed partial response (PR) per BICR and investigator according to RECIST v1.1.
Duration of Response As Assessed by Blinded Independent Central Review and Investigator Following I-DXd in Combination With Atezolizumab With Carboplatin (Part A and B of Cohort 2 Only) | From the date of first documentation of confirmed response (CR or PR) to the first documentation of objective progression or to death due to any cause, whichever occurs first, up to approximately 37 months
  Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (confirmed complete response [CR] or confirmed partial response [PR]) to the date of the first documentation of progressive disease (PD) or death due to any cause, whichever occurs first. The DoR will be calculated for responding participants (confirmed PR or confirmed CR) only.
Disease Control Rate As Assessed by Blinded Independent Central Review and Investigator Following I-DXd in Combination With Atezolizumab With Carboplatin (Part A and B of Cohort 2 Only) | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 37 months
  Disease control rate is defined as the proportion of participants who have achieved a best overall response of confirmed CR, confirmed PR, or SD by BICR and investigator assessment per RECIST v1.1.
Clinical Benefit Rate as Assessed by Blinded Independent Central Review and Investigator Following I-DXd in Combination With Atezolizumab With Carboplatin (Part A and B of Cohort 2 Only) | Baseline up until documented progressive disease, death, lost to follow-up, or withdrawal by the participant, up to approximately 37 months
  Clinical benefit rate (CBR) is defined as the proportion of participants who achieved a best overall response of confirmed CR, confirmed PR, or SD lasting for at least 180 days.
Time to Response As Assessed by Blinded Independent Central Review and Investigator Following I-DXd in Combination With Atezolizumab With Carboplatin (Part A and B of Cohort 2 Only) | From the start date of study drug to the date of the first documentation of response (CR or PR) that is subsequently confirmed, up to approximately 37 months
  Time to response (TTR) is defined as the time from the date of enrollment/randomization to the date of the first documentation of objective response (confirmed CR or confirmed PR) in responding subjects.
Best Percentage Change in the Sum of Diameters (SoD) of Measurable Tumors As Assessed by Blinded Independent Central Review and Investigator Following I-DXd in Combination With Atezolizumab With Carboplatin (Part A and B of Cohort 2 Only) | Baseline up to approximately 37 months
  The best percentage change in SoD is defined as the percentage change in the smallest SoD from all post-baseline tumor assessments, taking as reference the baseline SoD.
Overall Survival Following I-DXd in Combination With Atezolizumab With or Without Carboplatin (Part A and B) | From the start date of study drug to the date of death due to any cause, whichever occurs first, up to approximately 37 months
  Time from the date of enrollment/randomization to the date of death due to any cause.
Pharmacokinetic Parameter Maximum Serum Concentration of I-DXd | Cycle 1 Day 1 pre-dose up to Cycle 9 (and every 2 cycles thereafter up to 37 months) Day 1 pre-dose (each cycle is 21 days)
  Maximum serum concentration (Cmax) will be assessed using non-compartmental methods.
Pharmacokinetic Parameter Time to Maximum Serum Concentration of I-DXd | Cycle 1 Day 1 pre-dose up to Cycle 9 (and every 2 cycles thereafter up to 37 months) Day 1 pre-dose (each cycle is 21 days)
  Time to maximum serum concentration (Tmax) will be assessed using non-compartmental methods.
Pharmacokinetic Parameter Area Under the Concentration Curve of I-DXd | Cycle 1 Day 1 pre-dose up to Cycle 9 (and every 2 cycles thereafter up to 37 months) Day 1 pre-dose (each cycle is 21 days)
  Area under the concentration-time curve up to the last quantifiable time (AUClast) and Area under the concentration-time curve during dosing interval (AUCtau) will be assessed using non-compartmental methods.
The Number of Participants Who Are Anti-Drug Antibody (ADA)-Positive At Any Time and Who Have A Treatment-emergent Anti-Drug Antibody | Baseline up to approximately 37 months
  The ADA prevalence, which is the percentage of participants who are ADA positive at any time point (baseline or postbaseline), as well as the ADA incidence, which is the proportion of participants having treatment-emergent ADA during the study period, will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (58):
- United States (26):
  - University of Alabama -Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - David Geffen School of Medicine, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Advent Health Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Astera Cancer Care, East Brunswick, New Jersey
  - John Theurer Cancer Center At Hackensack Umc, Hackensack, New Jersey
  - New York University Cancer Center - Laura and Isaac Perlmutter Cancer Center At Nyu Langone, Mineola, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Hervert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - Lancaster General Hospital - Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital - Central, Philadelphia, Pennsylvania
  - Scri Oncology Partners, Nashville, Tennessee
  - Next Virginia, Fairfax, Virginia
  - Northwest Cancer Specialists, P.C.-Vancouver, Vancouver, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (9):
  - Hopital Albert Calmette - Chu Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital de la Timone, Marseille
  - Institut Curie - Site de Paris, Paris
  - Hopital Tenon, Paris
  - Chu Rennes - Hopital Pontchaillou, Rennes
  - CHU Nantes - Hôpital Guillaume et René Laënnec, Saint-Herblain
  - Hôpital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Japan (11):
  - NHO Himeji Medical Center, Himeji-shi
  - Kansai Medical University Hospital, Hirakata-shi
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of Jfcr, Kōtoku
  - Social Welfare Organization Saiseikai Imperial Gift Foundation, Inc. Saiseikai Kumamoto Hospital, Kumamoto
  - Shizuoka Cancer Center, Nagaizumi-cho
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Kindai University Hospital, Ōsaka-sayama
  - Tokushima University Hospital, Tokushima
  - Fujita Health University Hospital, Toyoake-shi
- Spain (12):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Ico Girona - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Next Madrid, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Alvaro Cunqueiro, Vigo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/